CLINICAL TRIAL: NCT00574886
Title: Pilot Trial for Idiotype Vaccine Following High-Dose Chemotherapy and Hematopoietic Stem Cell Transplantation for Patients With Lymphoma Who Had Failed Induction Chemotherapy
Brief Title: Idiotype Vaccine After Chemotherapy & Stem Cell Transplantation in Lymphoma With Failed Induction Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Genitope Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0267-00-FB
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- 1 High dose BEAM chemotherapy, transplant & idiotype vaccine therapy (Experimental): This is a compassionate use protocol for participants who failed induction chemotherapy + Vaccine on previous trials. These participants then went on to high dose BEAM chemotherapy and transplant, then received idiotype vaccine therapy at 3 months post transplant. Vaccine was given monthly x 4 series, with a fifth series given 12 weeks after the fourth. Participants were then followed annually until progression or death with standard staging.
  Interventions: Biological: Id-KLH

INTERVENTIONS:
Biological: Id-KLH — Idiotype vaccine - .5mg recombinant idiotype immunoglobulin protein given subcutaneously for a total of five administrations over 6 months.
  Other Names: Vacmun KLH

SUMMARY:
This is a compassionate use protocol for participants who failed induction chemotherapy + Vaccine on previous trials. These participants then went on to high dose BEAM chemotherapy and transplant, then received idiotype vaccine therapy at 3 months post transplant. Vaccine was given monthly x 4 series, with a fifth series given 12 weeks after the fourth. Participants were then followed annually until progression or death with standard staging.

DETAILED DESCRIPTION:
This trial was made available as a compassionate use protocol for participants who failed induction chemotherapy + Vaccine on trials 0197-99-FB and 0196-99-FB. These follicular NHL participants then went on to high dose BEAM chemotherapy and transplant. Patients received idiotype vaccine therapy at 3 months post transplant. Vaccine was given monthly x 4 series, with a fifth series given 12 weeks after the fourth. Participants are then followed annually until progression or death with standard staging. Immune response testing continues annually on participants who continue to have a response post transplant.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed aggressive or indolent, B-cell non-hodgkins lymphoma
* original enrollment in vaccine protocol for newly diagnosed lymphoma and had successful production of idiotype vaccine
* failed to achieve PR or CR with initial induction chemotherapy, received salvage chemotherapy and then stem cell transplant and achieved a CR or good PR following transplantation

  ->/= 19 years
* signed informed consent
* non-pregnant, non-lactating

Exclusion Criteria:

* serious disease or condition that, in the opinion of the investigator, would compromise the subject's ability to participate in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2000-08-03 (Actual); Primary Completion 2002-03-01 (Actual); Study Completion 2008-04-15 (Actual)

PRIMARY OUTCOMES:
Humoral and cellular responses to idiotype vaccine following high-dose chemotherapy and hematopoietic stem cell transplant | After vaccination
  Humoral and cellular responses to idiotype vaccine with KLH and GM-CSF adjuvant given to patients with lymphoma following high-dose chemotherapy and

SECONDARY OUTCOMES:
Safety and toxicity of idiotype vaccine post-transplant setting | Post-transplant vaccination
  Safety and toxicity of idiotype vaccine with KLH and GM-CSF adjuvant in the post-transplant setting

CONTACTS AND LOCATIONS:
Overall Officials: Julie Vose, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States